CLINICAL TRIAL: NCT06828276
Title: Culturally and Language-Adapted i-CBT for Common Mental Health Problems: A Randomized Controlled Study With Farsi/Dari-Speaking Migrants
Brief Title: Culturally Adapted i-CBT for Farsi/Dari Speaking Migrants
Acronym: i-CBT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Shervin Shahnavaz, PhD, Lecturer, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KI-CNS-20250117
Record Dates: First submitted 2025-01-22; First posted 2025-02-14 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: Depressive Symptoms; Anxiety Symptoms; Grief; Psychological Trauma; Insomnia; Resilience; Stress; Psychological Well Being; Marital Relationship; Wellbeing; Common Mental Health Problems; Rumination
Keywords: Refugee; Cognitive behavioral therapy; Psychological problems; Persian speaking; Psychological well-being; Youth; Mental problems; Resilience; Asylum seeker
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Trauma; Sleep Initiation and Maintenance Disorders; Psychological Well-Being; Rumination Syndrome

STUDY DESIGN:
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): Tailored I-CBT for mild to moderate common mental health problems over a 10-weeks-period.
  Interventions: Behavioral: Culturally adapted i-CBT
- Waiting-list (No Intervention): Control group

INTERVENTIONS:
Behavioral: Culturally adapted i-CBT — A culturally and language adapted i-CBT intervention for Farsi/Dari speaking youth migrants and refugees. The intervention targets mild to moderate common mental health problems.
  Arms: Active group

SUMMARY:
The aim of this randomized controlled trial (RCT) is to investigate the effectiveness of a culturally adapted internet-based cognitive behavioral therapy (i-CBT) intervention in reducing symptoms of common mental health issues among Farsi/Dari-speaking youth migrants and refugees. Investigator hypothesizes that there will be a significant decrease in psychological symptoms after participants receive the intervention compared to a control group.

DETAILED DESCRIPTION:
Participants who are included in the study will be allocated to the experimental group and the control group (waiting list). Participants will be invited to participate tailored i-CBT intervention over 10-weeks. Intervention covers common psychological issues. Participants will have access to support through a chatting function, during the interventional period. Intervention effects will be measured prior-treatment, post-treatment, and 6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 15 and 29.
* A score above the cut-off 1.75 on HSCL-25
* Has a refugee or migrant background
* Has a good and stable internet connection
* Has access to a computer, tablet or smartphone
* Is fluent in reading and writing Arabic
* Has the ability to dedicate time to take part in the intervention for 6-10 weeks.

Exclusion Criteria:

* Is suffering from a severe mental illness, such as psychosis or severe depression.
* Is suffering from substance abuse
* Is undergoing a psychological treatment
* Has a high risk of suicide

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Hopkins Symptom Checklist-25 (HSCL-25) | Pre-intervention, up to 5 weeks, immediately after the intervention, 6 months after completion of the intervention
  Assessment of anxiety and depressive symptoms. HSCL-25 consists of 25 items.Each item is rated on a scale from 1 to 4, where 1 means "Not at all" and 4 means "Extremely".Higher scores indicate a worse outcome, as they reflect greater severity of symptoms.

SECONDARY OUTCOMES:
Psychological Outcome Profiles (PSYCHLOPS) | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  Impact of problematic area on function. PSYCHLOPS questionnaire consists of 4 items. These items are designed to capture the patient's main problem, the impact of this problem on their daily life, and their overall well-being. Each question in PSYCHLOPS is scored on a scale from 0 to 5, where 0 indicates no problem and 5 indicates the most severe problem. Higher scores indicate a worse outcome, as they reflect greater severity of problems or distress.
Insomnia Severity Index (ISI) | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  Assessment of severity of insomnia symptoms. ISI consists of 7 items, each rated on a scale from 0 to 4.Higher scores indicate a worse outcome, as they reflect more severe insomnia symptoms.
Prolonged Grief Disorder (PG-13) | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  Assessment of prolonged grief disorder. The PG-13 consists of 13 items, each rated on a scale from 1 to 5, where 1 means "Not at all" and 5 means "Several times a day". Higher scores indicate a worse outcome, as they reflect more severe symptoms of prolonged grief.
Posttraumatic Stress Disorder Checklist (PCL-5) | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  Assessment of symptoms of post-traumatic stress disorder. The PCL-5 consists of 20 items, each rated on a scale from 0 to 4. The total score ranges from 0 to 80. Higher scores indicate a worse outcome, as they reflect greater severity of PTSD symptoms.
The World Health Organization-Five Well-Being Index (WHO-5) | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  Assessment of subjective psychological well-being.The WHO-5 consists of 5 items, each rated on a scale from 0 to 5. Higher scores indicate a better outcome, as they reflect higher levels of well-being.
Brief Resilience Scale (BRS) | Pre-intervention, immediately after the intervention, 6 months after completion of the intervention
  Assessment of resilience.The BRS consists of 6 items, each rated on a scale from 1 to 5. Higher scores indicate a better outcome, as they reflect greater resilience.
Client Satisfaction Questionnaire (CSQ-3) | Immediately after the intervention, 6 months after completion of the intervention
  Assessment of the levels of satisfaction of the participant with the intervention.CSQ-3 consists of 3 items. Each item is rated on a scale from 1 to 4. Higher scores indicate a better outcome, as they reflect greater satisfaction with the services received.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Background] Demetry Y, Wasteson E, Lindegaard T, Abuleil A, Geranmayeh A, Andersson G, Shahnavaz S. Individually Tailored and Culturally Adapted Internet-Based Cognitive Behavioral Therapy for Arabic-Speaking Youths With Mental Health Problems in Sweden: Qualitative Feasibility Study. JMIR Form Res. 2023 Nov 24;7:e46253. doi: 10.2196/46253. PMID 37999955
- [Background] Lindegaard T, Wasteson E, Demetry Y, Andersson G, Richards D, Shahnavaz S. Investigating the potential of a novel internet-based cognitive behavioural intervention for Dari and Farsi speaking refugee youth: A feasibility study. Internet Interv. 2022 Apr 1;28:100533. doi: 10.1016/j.invent.2022.100533. eCollection 2022 Apr. PMID 35433279
- See also: Description Registration page — http://rahafarsi.com
- See also: Description About the research project — https://liu.se/en/research/saha